CLINICAL TRIAL: NCT01924871
Title: Comparison of Deep Extubation During Emergence Using Desflurane or Desflurane With Remifentanil in Patients Undergoing General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Chongwha Baek, Chongwha Baek, MD, Ph.D, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: deep extubation in CAUH
Record Dates: First submitted 2013-08-12; First posted 2013-08-19 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Deep Extubation
MeSH Terms: interventions — Desflurane; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Desflurane group (Active Comparator): 1.5 MAC desflurane until extubation
  Interventions: Drug: Desflurane
- Desflurane with remifentanil group (Active Comparator): 1.0 MAC desflurane with 1.0ng/ml targeted concentration infusion of remifentanil
  Interventions: Drug: Desflurane with remifentanil

INTERVENTIONS:
Drug: Desflurane with remifentanil — During the emergence from anesthesia,extubation was performed under 1.0 MAC desflurane with 1.0ng/ml remifentanil
  Other Names: desflurane with remifetanil group
  Arms: Desflurane with remifentanil group
Drug: Desflurane — During the emergence from anesthesia,extubation was performed under 1.5 MAC desflurane
  Other Names: Desflurane alone group
  Arms: Desflurane group

SUMMARY:
It has been reported that deep extubation can reduce cardiopulmonary complication against endotracheal tube extubation during emergence from general anesthesia. The investigators hypothesized that using desflurane with target controlled infusion of remifentanil is more effective than using desflurane alone during deep extubation. The purpose of this study is to evaluate the effect of remifentanil to prevent respiratory complication (etc. coughing) during emergence from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60
* patients undergoing elective surgery take more than an hour
* Under general anesthesia using an LMA
* ASA I,II

Exclusion Criteria:

* Patients on CNS depressants
* Chronic opioid use
* Corticosteroid
* Pregnant patients
* Full stomach
* Morbidly obese (BMI >35kg/m2)
* Hepatitis B
* Hepatitis C
* Coronary artery disease
* Liver disease
* Renal disease
* Seizure disorder

Dropout criteria:

* Need for reintubation due to breath holding
* high ETCO2 during self ventilation (ETCO2>50)
* Surgeon or patient request

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desflurane Group | Desflurane With Remifentanil Group
Started | 31 | 31
Completed | 25 | 29
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desflurane Group | Desflurane With Remifentanil Group | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.76 (11.53) | 43.24 (9.39) | 42.17 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Awakening Time
Description: The outcomes assessor will record from the time of extubation in operating room to the time of eye opening and mouth opening
Time Frame: Participants will be followed from the time of extubation in operating room to the time of discharge from recovery room, an expected average of 1day.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Desflurane Group | Desflurane With Remifentanil Group
Number analyzed (Participants) | 25 | 29
minutes | 10 [8.5 to 10.5] | 7 [6 to 8]

2. Secondary Outcome: Success Rate & Complication Rate Including Cough
Description: We will assess the success rate of deep extubation without complication and the occurrence of cough during emergence from general anesthesia.
Time Frame: assessing the success rate of deep extubation without complication and the occurrance of cough from the completion of surgery to 5minute after extubation.
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Postoperative Pain
Description: The outcomes assessor will evaluate the degree of postoperative pain using a numeric rating scale (NRS). (0 = no pain, 10 = unimaginable severe pain)
Time Frame: Participants will be followed for the duration of postanesthesia care unit (PACU) stay, an expected average of 1 hour.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Desflurane Group | Desflurane With Remifentanil Group
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No